CLINICAL TRIAL: NCT03345082
Title: A Dose-Ranging Study of Intravitreal OPT-302 in Combination With Ranibizumab, Compared With Ranibizumab Alone, in Participants With Neovascular Age-Related Macular Degeneration (Wet AMD)
Brief Title: A Dose Ranging Study of OPT-302 With Ranibizumab in Neovascular (Wet) AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Opthea Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPT-302-1002
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-01

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.5 mg ranibizumab with 2.0 mg OPT-302 (Experimental): 0.5 mg ranibizumab intravitreal injection (0.05 ml) followed by 2.0 mg OPT-302 intravitreal injection (0.05 ml)
  Interventions: Biological: OPT-302; Biological: ranibizumab
- 0.5 mg ranibizumab with 0.5 mg OPT-302 (Experimental): 0.5 mg ranibizumab intravitreal injection (0.05 ml) followed by 0.5 mg OPT-302 intravitreal injection (0.05 ml)
  Interventions: Biological: OPT-302; Biological: ranibizumab
- 0.5 mg ranibizumab with sham (Sham Comparator): 0.5 mg ranibizumab intravitreal injection (0.05 ml) followed by sham
  Interventions: Biological: ranibizumab; Other: sham intravitreal injection

INTERVENTIONS:
Biological: OPT-302 — Intravitreal injection
  Arms: 0.5 mg ranibizumab with 0.5 mg OPT-302; 0.5 mg ranibizumab with 2.0 mg OPT-302
Biological: ranibizumab — Intravitreal injection
  Other Names: Lucentis
Other: sham intravitreal injection — Sham (mock) intravitreal injection
  Arms: 0.5 mg ranibizumab with sham

SUMMARY:
A multicentre, randomised, parallel group, sham-controlled, double-masked, dose-ranging study, investigating two doses of OPT-302 in combination with ranibizumab compared with ranibizumab with sham, over six consecutive monthly dosing cycles in participants with neovascular (wet) AMD.

ELIGIBILITY:
Inclusion Criteria:

* Active subfoveal choroidal neovascular (CNV) lesion or juxtafoveal lesion secondary to age-related macular AMD
* An ETDRS BCVA score between 60 and 25 (inclusive) letters

Exclusion Criteria:

* Previous treatment for wet AMD or previous treatment for CNV due to other causes in the Study Eye
* Clinically significant ocular disorders which may interfere with assessment of visual acuity, assessment of toxicity, or fundus photography in the Study Eye
* Poorly controlled diabetes mellitus (defined as HbA1c>7%)
* Any clinically significant cardiovascular, renal or hepatic conditions, recent surgery, or malignancy, that would make the participant unsuitable for the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
Mean change in Early Treatment Diabetic Retinopathy Study (ETDRS) best corrected visual acuity (BCVA) | Baseline to Week 24

SECONDARY OUTCOMES:
Proportion of participants gaining 15 or more ETDRS BCVA letters | Baseline to Week 24
Area under the ETDRS BCVA over time curve | Baseline to Week 24
Change in central subfield thickness (CST) on spectral domain optical coherence tomography (SD-OCT) | Baseline to Week 24
Change in intra-retinal fluid and sub-retinal fluid on SD-OCT | Baseline to Week 24
Proportion of participants losing 15 or more letters (on ETDRS BCVA chart) | Baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Opthea Limited
Locations (97):
- United States (53):
  - Opthea Investigational Site, Phoenix, Arizona
  - Opthea Investigational Site, Beverly Hills, California
  - Opthea Investigational Site, Encino, California
  - Opthea Investigational Site, Palm Desert, California
  - Opthea Investigational Site, Redlands, California
  - Opthea Study Site, Sacramento, California
  - Opthea Investigational Site, Sacramento, California
  - Opthea Investigational Site, San Diego, California
  - Opthea Investigational Site, Santa Ana, California
  - Opthea Investigational Site, Santa Barbara, California
  - Opthea Investigational Site, Santa Maria, California
  - Opthea Investigational Site, Colorado Springs, Colorado
  - Opthea Investigational Site, Golden, Colorado
  - Opthea Investigational Site, Boynton Beach, Florida
  - Opthea Investigational Site, Fort Myers, Florida
  - Opthea Investigational Site, Melbourne, Florida
  - Opthea Investigational Site, Pensacola, Florida
  - Opthea Investigational Site, St. Petersburg, Florida
  - Opthea Investigational Site, Tallahassee, Florida
  - Opthea Investigational Site, Winter Haven, Florida
  - Opthea Investigational Site, Augusta, Georgia
  - Opthea Investigational Site, Shawnee Mission, Kansas
  - Opthea Investigational Site, Wichita, Kansas
  - Opthea Investigational Site, Paducah, Kentucky
  - Opthea Investigational Site, Baltimore, Maryland
  - Opthea Investigational Site, Grand Rapids, Michigan
  - Opthea Investigational Site, Las Vegas, Nevada
  - Opthea Investigational Site, Reno, Nevada
  - Opthea Investigational Site, Edison, New Jersey
  - Opthea Investigational Site, Teaneck, New Jersey
  - Opthea Investigational Site, Albuquerque, New Mexico
  - Opthea Investigational Site, Lynbrook, New York
  - Opthea Investigational Site, Rochester, New York
  - Opthea Investigational Site, Syracuse, New York
  - Opthea Investigational Site, Asheville, North Carolina
  - Opthea Investigational Site, Charlotte, North Carolina
  - Opthea Investigational Site, Cleveland, Ohio
  - Opthea Investigational Site, Columbus, Ohio
  - Opthea Investigational Site, Portland, Oregon
  - Opthea Investigational Site, Camp Hill, Pennsylvania
  - Opthea Investigational Site, Kingston, Pennsylvania
  - Opthea Investigational Site, Philadelphia, Pennsylvania
  - Opthea Investigational Site, Ladson, South Carolina
  - Opthea Investigational Site, West Columbia, South Carolina
  - Opthea Investigational Site, Abilene, Texas
  - Opthea Investigational Site, Austin, Texas
  - Opthea Investigational Site, Houston, Texas
  - Opthea Investigational Site, San Antonio, Texas
  - Opthea Investigational Site, The Woodlands, Texas
  - Opthea Investigational Site, Willow Park, Texas
  - Opthea Investigational Site, Fairfax, Virginia
  - Opthea Investigational Site, Virginia Beach, Virginia
  - Opthea Investigational Site, Silverdale, Washington
- Czechia (2):
  - Opthea Investigational Site, Hradec Králové
  - Opthea Investigational Site, Prague
- France (5):
  - Opthea Investigational Site, Créteil
  - Opthea Investigational Site, Dijon
  - Opthea Investigational Site, Écully
  - Opthea Investigational Site, Paris
  - Opthea Investigational Site, Strasbourg
- Hungary (3):
  - Opthea Investigational Site, Budapest
  - Opthea Investigational Site, Nyíregyháza
  - Opthea Investigational Site, Szeged
- Israel (6):
  - Opthea Investigational Site, Haifa
  - Opthea Investigational Site, Jerusalem
  - Opthea Investigational Site, Kfar Saba
  - Opthea Investigational Site, Petah Tikva
  - Opthea Investigational Site, Rehovot
  - Opthea Investigational Site, Tel Aviv
- Italy (4):
  - Opthea Investigational Site, Bologna
  - Opthea Investigational Site, Florence
  - Opthea Investigational Site, Milan
  - Opthea Investigational Site, Roma
- Latvia (2):
  - Opthea Investigational Site, Jelgava
  - Opthea Investigational Site, Riga
- Poland (7):
  - Opthea Investigational Site, Bydgoszcz
  - Opthea Investigational Site, Gdansk
  - Opthea Investigational Site, Katowice
  - Opthea Investigational Site, Krakow
  - Opthea Investigationa Site, Lublin
  - Opthea Investigational Site, Lublin
  - Opthea Investigational Site, Wroclaw
- Spain (8):
  - Opthea Investigational Site, Barcelona
  - Opthea Investigational Site, Bilbao
  - Opthea Investigational Site, Madrid
  - Opthea Investigational Site, Oviedo
  - Opthea Investigational Site, Pamplona
  - Opthea Investigational Site, Santiago de Compostela
  - Opthea Investigational Site, Valencia
  - Opthea Investigational Site, Valladolid
- United Kingdom (7):
  - Opthea Investigational Site, Bristol
  - Opthea Investigational Site, Frimley
  - Opthea Investigational Site, Glasgow
  - Opthea Investigational Site, London
  - Opthea Investigational Site, Maidstone
  - Opthea Investigational Site, Sheffield
  - Opthea Investigational Site, Wolverhampton

REFERENCES:
- [Derived] Jackson TL, Slakter J, Buyse M, Wang K, Dugel PU, Wykoff CC, Boyer DS, Gerometta M, Baldwin ME, Price CF; Opthea Study Group Investigators. A Randomized Controlled Trial of OPT-302, a VEGF-C/D Inhibitor for Neovascular Age-Related Macular Degeneration. Ophthalmology. 2023 Jun;130(6):588-597. doi: 10.1016/j.ophtha.2023.02.001. Epub 2023 Feb 6. PMID 36754174